CLINICAL TRIAL: NCT06683729
Title: HighLife Clarity Treatment of Severe Mitral Regurgitation
Acronym: HIGHFIVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HighLife SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-2024-01-Pivotal
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Mitral Valve (MV) Regurgitation
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single-arm study (Experimental): Single-arm, group sequential, prospective, multicenter, global, open-label study for the investigation of the safety and effectiveness of the HighLife transcatheter trans-septal mitral valve replacement (SMVR) System. The HighLife TSMVR system is intended for use for percutaneous mitral valve replacement via trans-septal access in patients suffering from symptomatic moderate-to-severe or severe functional (secondary) mitral regurgitation (MR).
  Interventions: Device: Trans-septal (TS) Mitral Valve Replacement (TSMVR) Valve system

INTERVENTIONS:
Device: Trans-septal (TS) Mitral Valve Replacement (TSMVR) Valve system — Trans-catheter, trans-septal mitral valve replacement.

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the HighLife transcatheter trans-septal mitral valve replacement (TSMVR) system in NYHA Class ≥ II-IV patients with moderate-to-severe or severe mitral regurgitation (MR) who, by assessment of the local Heart Team, are unsuitable for treatment with approved transcatheter repair (sub-optimal results to complex or prohibitive edge-to-edge repair) or surgical mitral valve intervention according to guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Based on local regulations, the subject meets the legal minimum age to provide informed consent
* Moderate-to-severe or severe symptomatic MR (≥3+) by transthoracic echocardiography (TTE) which is primarily due to lack of mitral leaflet coaptation, secondary to either a) LV cardiomyopathy with restriction of the mitral leaflet(s), or b) mitral annular dilatation due to chronic atrial fibrillation or other cause, as confirmed by the echocardiographic core laboratory (note: some element of primary (degenerative) MR may be present, but the core lab must agree that the principal etiology is secondary MR)
* New York Heart Association (NYHA) functional class II, III or ambulatory IV
* Based on the assessment of the local multidisciplinary heart team, the patient is:

  1. being treated with stable maximally-tolerated doses of guidelines class I indicated GDMT for at least one month, and CRT for at least 3 months (if applicable)
  2. not indicated for heart surgery (mitral valve repair or replacement) according to guidelines and the local standard of care
  3. unsuitable for treatment with transcatheter edge-to-edge repair (complex TEER anatomy) as assessed by the site interventional cardiologist(s)

Exclusion Criteria:

* Any stroke or TIA within 30 days prior to procedure; any prior intracranial hemorrhage at any time; or any intracerebral mass, arteriovenous fistula or other malformation or defect predisposing to bleeding
* Known severe carotid stenosis (>70% diameter stenosis by non-invasive imaging) or carotid stenting or carotid endarterectomy within 30 days)
* History of bleeding diathesis, coagulopathy, clotting disorder, or refusal of future blood transfusion or bleeding in the 3 months prior to procedure other than minor cutaneous bleeding
* Patients in whom transesophageal echo (TEE) is not feasible
* Chronic obstructive pulmonary disease (COPD) requiring continuous home oxygen therapy or chronic outpatient oral steroid use.
* Female subjects of childbearing potential who are not willing or able to comply with the use of contraception, or who are pregnant or lactating, or plan to get pregnant within the next 12 months.
* Participation in another clinical study of an investigational drug or device at the time of inclusion that has not reached its primary endpoint
* Patient has known allergies to the device components or contrast medium, which cannot be medically managed
* Patient cannot tolerate anticoagulation (i.e. warfarin), or not willing to take anticoagulation for at least 6 months, or antiplatelet agents (i.e. aspirin, clopidogrel)
* Patient with a life expectancy of less than 12 months, or otherwise is unable to comply with the follow-up schedule and assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality or heart failure (HF) hospitalization | 24 months
  The rate of all-cause mortality or heart failure (HF) hospitalization at 24 months post-implant.